CLINICAL TRIAL: NCT06730737
Title: Brief Lifestyle Medicine Preventive Randomized Prospective Interactive Educational Intervention in the Primary Care Clinic
Brief Title: Lifewise Preventive Video Education in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health-Livonia (Other)
Responsible Party: Principal Investigator, Daniel Keyes, MD, MPH, Associate Chair, Academic Affairs, Principal Investigator, Trinity Health-Livonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TrinityHealthLivonia
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Prevention Harmful Effects; Health Maintenance; Preventive Health Care; Dietary Habits
Keywords: Prevention; Lifestyle; coronary artery disease; video; video education; video education for adults; preventive health care
MeSH Terms: conditions — Feeding Behavior; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial of Interactive Preventive Video Education
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video intervention group (Experimental): The intervention is an interactive preventive education video lasting approximately 10 minutes. The video is interactive because it asks the patients to answer simple questions about the content in the video to keep them engaged. For instance, if the participant indicates that they do not smoke, the video will "skip" the smoking cessation education and move directly to the other prevention domains.
  Interventions: Other: Video preventive education
- Control (No Intervention): This arm consists of those randomized to receive no video

INTERVENTIONS:
Other: Video preventive education — Interactive video that teaches the subject about the overall importance of prevention, smoking cessation, proper diet, exercise, and sleep.
  Arms: Video intervention group

SUMMARY:
It is widely accepted that prevention is far more impactful than curative medicine and must be included in primary care. In a previous pilot study, we evaluated passive video preventive lifestyle education in the emergency department. The current study is a randomized prospective trial assessing the practicality and impact of a brief interactive educational video intervention to patients during primary care clinic visits.

DETAILED DESCRIPTION:
Background and Summary of Objectives: It is widely accepted that prevention is far more impactful than curative medicine concerning overall health efficacy. The primary care setting faces the challenges of increasingly important time constraints and conflicting priorities. However, prevention is a priority regarding the improvement in health outcomes. In a previous pilot study, we investigated the impact of a simple instructional video on patients' willingness to change in the emergency department setting. The initial intervention was passive, requiring subjects to watch a video without interaction. The current study evaluates the practicality and impact of bringing a brief interactive educational video intervention to patients at the primary care clinic visit.

Summary of Study Design This randomized, non-blinded prospective study of "just in time" education for adult patients presenting to the primary care clinic immediately following their primary care appointment.

Patients will be randomized to receive the interactive intervention video during this encounter with the practitioner in the clinic. The intervention is an interactive video with a duration of approximately 10-15 minutes. The video is interactive because it asks the patients to answer simple questions about the content in the video to keep them engaged with the content. For instance, if the participant indicates that they do not smoke, the video will "skip" the smoking cessation education and move directly to the other prevention domains. Before leaving the clinic, all patients will be presented with a questionnaire about their readiness and confidence to initiate lifestyle changes (transtheoretical stage of change measured on a "readiness ruler") and additional survey instruments. Most of these questions will come from existing validated scales, including the Gillespie & Lenz behavior modification tool, the Pittsburgh Sleep Quality Index, and select questions from the US HCAHPS Patient Satisfaction Survey. They will be asked for access to their medical record and their willingness to be contacted for a follow-up survey.

Outcome measures:

The study's primary outcome will be the results of the Lifestyle Readiness to Change and Confidence to Change questionnaires. Secondary outcomes will include satisfaction with the primary care clinic visit using select questions from HCAHPS, and whether they intend to change any specific lifestyle behavior (dichotomous, yes/no) and, if yes, to specific which one(s), seeking medical care outside of the clinic visit as determined by a review of the patient's medical record at intervals of 30 days and six months. HIV will not be evaluated outside of its inclusion in the Charlson Comorbidity Index (CCI). A follow-up survey at approximately 3-12 months will evaluate new diagnoses related to chest pain and ask about the individual's lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 80, inclusive.

Exclusion Criteria:

* Non-English-speaking patient
* Unable or unwilling to consent to the study
* Unable or unwilling to hear a video on a smartphone or computer tablet
* The patient is in hospice care
* Patients with advanced dementia, in the opinion of the person administering the survey

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Lifestyle Readiness to Change and Confidence to Change questionnaires | Immediately following exposure to the intervention or not (both arms receive the questionnaires)
  The study's primary outcome will be the results of the Lifestyle Readiness to Change and Confidence to Change questionnaires.

SECONDARY OUTCOMES:
Satisfaction, intent to changve lifestyle behavior, follow up clinic visit | 18 months
  satisfaction with the primary care clinic visit using select questions from HCAHPS, and whether they intend to change any specific lifestyle behavior (dichotomous, yes/no) and, if yes, to specific which one(s), seeking medical care outside of the clinic visit as determined by a review of the patient's medical record within approximately six months. A follow-up survey at approximately 3-12 months will evaluate new diagnoses related to chest pain and ask about the individual's lifestyle changes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keyes, MD, MPH, Principal Investigator — Trinity Health-Livonia
Locations (1):
- Trinity Health-Livonia Hospital and Affiliated Clinics, Livonia, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The data contains patient health information (PHI), and currently, there is no plan for public disclosure of the data.

REFERENCES:
- [Background] Wood EB, Harrison G, Trickey A, Friesen MA, Stinson S, Rovelli E, McReynolds S, Presgrave K. Evidence-Based Practice: Video-Discharge Instructions in the Pediatric Emergency Department. J Emerg Nurs. 2017 Jul;43(4):316-321. doi: 10.1016/j.jen.2016.11.003. Epub 2017 Mar 28. PMID 28359707
- [Background] Stange KC, Flocke SA, Goodwin MA, Kelly RB, Zyzanski SJ. Direct observation of rates of preventive service delivery in community family practice. Prev Med. 2000 Aug;31(2 Pt 1):167-76. doi: 10.1006/pmed.2000.0700. PMID 10938218
- [Background] Schuling J, de Haan R, Limburg M, Groenier KH. The Frenchay Activities Index. Assessment of functional status in stroke patients. Stroke. 1993 Aug;24(8):1173-7. doi: 10.1161/01.str.24.8.1173. PMID 8342192
- [Background] Rising KL, Padrez KA, O'Brien M, Hollander JE, Carr BG, Shea JA. Return visits to the emergency department: the patient perspective. Ann Emerg Med. 2015 Apr;65(4):377-386.e3. doi: 10.1016/j.annemergmed.2014.07.015. Epub 2014 Aug 27. PMID 25193597
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Prochaska JO, DiClemente CC. Stages of change in the modification of problem behaviors. Prog Behav Modif. 1992;28:183-218. No abstract available. PMID 1620663
- [Background] Pickens GT, Moore B, Smith MW, McDermott KW, Mummert A, Karaca Z. Methods for estimating the cost of treat-and-release emergency department visits. Health Serv Res. 2021 Oct;56(5):953-961. doi: 10.1111/1475-6773.13709. Epub 2021 Aug 5. PMID 34350589
- [Background] Pathak S, Summerville G, Kaplan CP, Nouri SS, Karliner LS. Patient-Reported Use of the After Visit Summary in a Primary Care Internal Medicine Practice. J Patient Exp. 2020 Oct;7(5):703-707. doi: 10.1177/2374373519879286. Epub 2019 Oct 4. PMID 33294604
- [Background] Park H, Roubal AM, Jovaag A, Gennuso KP, Catlin BB. Relative Contributions of a Set of Health Factors to Selected Health Outcomes. Am J Prev Med. 2015 Dec;49(6):961-9. doi: 10.1016/j.amepre.2015.07.016. PMID 26590942
- [Background] Papa L, Seaberg DC, Rees E, Ferguson K, Stair R, Goldfeder B, Meurer D. Does a waiting room video about what to expect during an emergency department visit improve patient satisfaction? CJEM. 2008 Jul;10(4):347-54. doi: 10.1017/s1481803500010356. PMID 18652727
- [Background] McCarthy DM, Engel KG, Buckley BA, Huang A, Acosta F, Stancati J, Schmidt MJ, Adams JG, Cameron KA. Talk-time in the emergency department: duration of patient-provider conversations during an emergency department visit. J Emerg Med. 2014 Nov;47(5):513-9. doi: 10.1016/j.jemermed.2014.06.056. Epub 2014 Sep 8. PMID 25214177
- [Background] Hood CM, Gennuso KP, Swain GR, Catlin BB. County Health Rankings: Relationships Between Determinant Factors and Health Outcomes. Am J Prev Med. 2016 Feb;50(2):129-35. doi: 10.1016/j.amepre.2015.08.024. Epub 2015 Oct 31. PMID 26526164
- [Background] Hirabayashi KJ, Pomerantz M, Radell JE, Chadha N, Thomas S, Serle JB. The Efficacy of the After-visit Summary in Medication Recall Among Glaucoma Patients. J Glaucoma. 2020 Jul;29(7):529-535. doi: 10.1097/IJG.0000000000001518. PMID 32332333
- [Background] Goodacre R, Karim A, Kaderbhai MA, Kell DB. Rapid and quantitative analysis of recombinant protein expression using pyrolysis mass spectrometry and artificial neural networks: application to mammalian cytochrome b5 in Escherichia coli. J Biotechnol. 1994 May 15;34(2):185-93. doi: 10.1016/0168-1656(94)90088-4. PMID 7764850
- [Background] Colby SM, Monti PM, O'Leary Tevyaw T, Barnett NP, Spirito A, Rohsenow DJ, Riggs S, Lewander W. Brief motivational intervention for adolescent smokers in medical settings. Addict Behav. 2005 Jun;30(5):865-74. doi: 10.1016/j.addbeh.2004.10.001. Epub 2004 Nov 10. PMID 15893085
- [Background] Dhawan N, Saeed O, Gupta V, Desai R, Ku M, Bhoi S, Verma S. Utilizing video on myocardial infarction as a health educational intervention in patient waiting areas of the developing world: A study at the emergency department of a major tertiary care hospital in India. Int Arch Med. 2008 Jul 29;1(1):14. doi: 10.1186/1755-7682-1-14. PMID 18662408
- [Background] Ding R, McCarthy ML, Desmond JS, Lee JS, Aronsky D, Zeger SL. Characterizing waiting room time, treatment time, and boarding time in the emergency department using quantile regression. Acad Emerg Med. 2010 Aug;17(8):813-23. doi: 10.1111/j.1553-2712.2010.00812.x. PMID 20670318
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771